CLINICAL TRIAL: NCT05867901
Title: Clinical Research of Drug Holiday Based on MRD Detection in Gastrointestinal Stromal Tumor Patients at High Risk of Recurrence
Brief Title: Clinical Research of Drug Holiday Based on MRD Detection in GIST Patients at High Risk of Recurrence
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhidong Gao, Associate Clinical Professor of Department of Gastrointestinal Surgery, Peking University People's Hospital
Other Study IDs: 2023-076
Record Dates: First submitted 2023-04-23; First posted 2023-05-22 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Drug Holiday; Minimal Residual Disease; Circulating Tumor DNA
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissues and peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients cohort: As an one-arm observational clinical trial, we have only one patients cohort.

SUMMARY:
This study is aimed:

* to evaluate the dynamic monitoring value of MRD detection for postoperative recurrence in high-risk GIST patients;

  * to evaluate the effect of drug holiday mode based on MRD detection on progression-free Survival (PFS) and/or overall survival (OS) after drug withdrawal for high-risk GIST patients who have achieved disease control after long-term use of imatinib; ③ to investigate the response rate of imatinib re-use in patients who developed disease progression after drug withdrawal; ④ to explore whether the "drug holiday" treatment mode based on MRD detection could delay the occurrence of secondary imatinib resistance mutations for high-risk GIST patients with long-term use of imatinib after surgery.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) is the most common mesenchymal tumor of the gastrointestinal tract, and surgery is the preferred treatment method for primary resectable GIST. The guidelines recommend that patients at high risk of recurrence should be treated with tyrosine kinase inhibitors (TKI) such as imatinib for at least 3 years after surgery. However, in actual clinical practice, some patients face the situation of early withdrawal or prolonged medication, so the timing of drug withdrawal needs to be further studied. Recent studies have reported that some GIST patients who have achieved disease control through long-term use of imatinib can still achieve a long progression-free survival after drug withdrawal, and those who relapse after drug withdrawal can still achieve disease control after re-use of imatinib. This suggests that for some selected patients, a "drug holiday" treatment mode could be possible, in which drugs are discontinued when appropriate and restarted if necessary. How to select patients suitable for this mode of treatment needs further exploration. Liquid biopsy of peripheral blood circulating tumor DNA (ctDNA) to detect minimal residual disease (MRD) can be used for the diagnosis, efficacy evaluation, recurrence and drug resistance monitoring of a variety of malignant tumors. Existing studies have explored the "drug holiday" treatment mode based on MRD detection assisting patients with advanced non-small cell lung cancer to use TKI. Therefore, this one-arm prospective observational clinical study will assist some high-risk GIST patients who have been treated with imatinib for 3 years after surgery and have achieved disease control to adopt the treatment mode of "drug holiday" based MRD detection, aiming to evaluate the value of MRD detection in monitoring postoperative recurrence of high-risk GIST, investigate the effect of "drug holiday" treatment mode based on MRD detection on disease recurrence and patient survival, and to explore whether it can delay the occurrence of drug-resistant mutations.

ELIGIBILITY:
Inclusion Criteria:

* ① Age: ≥18 years and ≤75 years;
* ② The primary lesion (and metastatic lesion) underwent R0 or R1 surgical resection, and patients were clinically diagnosed with high recurrence risk GIST combined with postoperative pathological results;
* ③ The patient have received imatinib adjuvant therapy for 3 years after surgery, and no gross lesions were detected by imaging examination, and the possibility of drug withdrawal was considered based on the comprehensive judgment of the doctor in charge;
* ④ The liquid biopsy for baseline ctDNA is negative;
* ⑤ Primary Imatinib resistant mutations were not detected by genetic testing, such as SDH-deficient GIST, NF1-mutant GIST, BRAF-mutant GIST and GIST with NTRK3 rearrangement;
* ⑥ PS score is 0-1 and expected survival time is more than 4 months;
* ⑦ Patients are willing to stop drug use and observe, and patients and their families could understand the study protocol and voluntarily participate in this study, and signed informed consent. In the follow-up study, they could provide the clinical pathological data and imaging data needed for the study process, cooperate with the follow-up and collect the blood of the clinical efficacy evaluation, and agree to use the test data for the follow-up study and product development.

Exclusion Criteria:

* ① Fresh or paraffin tissue of the surgical tumor is not available;
* ② Not receiving the assigned treatment or change therapy before disease progression;
* ③ Unable to cooperate with follow-up with the study according to defined clinical period;
* ④ Unable to take or provide defined imaging assessment examinations;
* ⑤ Other conditions that investigators consider inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk GIST patients who have been treated with imatinib for more than 3 years after surgery and have no gross lesions in imaging examination
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progress-free Survival | From date when patients first enter the drug holiday until the date of imaging examinations confirmed disease progression up to 3 years
  Progression-free survival after patients first enter the drug holiday
Drug re-use rate | 3 years from the time when patients first enter the drug holiday
  The proportion of patients who take drug re-use due to disease progression within 3 years after first entering drug holiday
Drug retreatment response rate | 3 years from the time when patients first enter the drug holiday
  Drug response rate among patients who take drug re-use due to disease progression within 3 years after first entering drug holiday

SECONDARY OUTCOMES:
Overall Survival | From date when patients first enter the drug holiday until the date of death up to 3 years
  Overall survival after patients first enter the drug holiday
genetic mutation profiling of ctDNA-MRD | 3 years from the time when patients first enter the drug holiday
  Results of genetic mutations in patients after the conversion of MRD from negative to positive, especially the detection of secondary imatinib resistance mutations
MRD versus imaging examination | 3 years from the time when patients first enter the drug holiday
  compare the time of MRD conversion and the time of disease progression assessed by imaging examination

CONTACTS AND LOCATIONS:
Overall Officials: Zhidong Gao, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Begum FA, Rahman MA, Rabbi H, Mostofa G, Chowdhury Q. Primary Jejunal Gastrointestinal Stromal Tumor: Diagnosis Delay of 3 Years but Successful Management in Early Stage (II) by Surgery and Adjuvant Therapy. Gastrointest Tumors. 2019 Aug;6(1-2):36-42. doi: 10.1159/000496973. Epub 2019 Apr 3. PMID 31602375
- [Result] Mazur MT, Clark HB. Gastric stromal tumors. Reappraisal of histogenesis. Am J Surg Pathol. 1983 Sep;7(6):507-19. doi: 10.1097/00000478-198309000-00001. PMID 6625048
- [Result] Joensuu H. Risk stratification of patients diagnosed with gastrointestinal stromal tumor. Hum Pathol. 2008 Oct;39(10):1411-9. doi: 10.1016/j.humpath.2008.06.025. PMID 18774375
- [Result] Joensuu H, Eriksson M, Sundby Hall K, Reichardt A, Hermes B, Schutte J, Cameron S, Hohenberger P, Jost PJ, Al-Batran SE, Lindner LH, Bauer S, Wardelmann E, Nilsson B, Kallio R, Jaakkola P, Junnila J, Alvegard T, Reichardt P. Survival Outcomes Associated With 3 Years vs 1 Year of Adjuvant Imatinib for Patients With High-Risk Gastrointestinal Stromal Tumors: An Analysis of a Randomized Clinical Trial After 10-Year Follow-up. JAMA Oncol. 2020 Aug 1;6(8):1241-1246. doi: 10.1001/jamaoncol.2020.2091. PMID 32469385
- [Result] Joensuu H, Eriksson M, Sundby Hall K, Hartmann JT, Pink D, Schutte J, Ramadori G, Hohenberger P, Duyster J, Al-Batran SE, Schlemmer M, Bauer S, Wardelmann E, Sarlomo-Rikala M, Nilsson B, Sihto H, Monge OR, Bono P, Kallio R, Vehtari A, Leinonen M, Alvegard T, Reichardt P. One vs three years of adjuvant imatinib for operable gastrointestinal stromal tumor: a randomized trial. JAMA. 2012 Mar 28;307(12):1265-72. doi: 10.1001/jama.2012.347. PMID 22453568
- [Result] Raut CP, Espat NJ, Maki RG, Araujo DM, Trent J, Williams TF, Purkayastha DD, DeMatteo RP. Efficacy and Tolerability of 5-Year Adjuvant Imatinib Treatment for Patients With Resected Intermediate- or High-Risk Primary Gastrointestinal Stromal Tumor: The PERSIST-5 Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):e184060. doi: 10.1001/jamaoncol.2018.4060. Epub 2018 Dec 13. PMID 30383140
- [Result] Kang YK, Kim HD, Kim HJ, Park YS, Beck MY, Ryu MH. Interruption of imatinib in advanced gastrointestinal stromal tumor after prolonged imatinib maintenance in the absence of gross tumor lesions. Gastric Cancer. 2023 Jul;26(4):604-613. doi: 10.1007/s10120-023-01377-2. Epub 2023 Mar 8. PMID 36884149
- [Result] Howland RH. Medication holidays. J Psychosoc Nurs Ment Health Serv. 2009 Sep;47(9):15-8. doi: 10.3928/02793695-20090804-01. PMID 19772246
- [Result] Mouliere F, Thierry AR. The importance of examining the proportion of circulating DNA originating from tumor, microenvironment and normal cells in colorectal cancer patients. Expert Opin Biol Ther. 2012 Jun;12 Suppl 1:S209-15. doi: 10.1517/14712598.2012.688023. Epub 2012 May 18. PMID 22594497
- [Result] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Result] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Result] Mitchell SM, Ho T, Brown GS, Baker RT, Thomas ML, McEvoy A, Xu ZZ, Ross JP, Lockett TJ, Young GP, LaPointe LC, Pedersen SK, Molloy PL. Evaluation of Methylation Biomarkers for Detection of Circulating Tumor DNA and Application to Colorectal Cancer. Genes (Basel). 2016 Dec 15;7(12):125. doi: 10.3390/genes7120125. PMID 27983717
- [Result] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368